Republic of Iraq
Ministry of Higher Education
and scientific Research
University of Baghdad
College of Dentistry



## Efficacy of C-PRF versus I-PRF on gingival thickness & keratinized tissue width in subjects with thin gingival biotype: (Split Mouth Controlled Clinical Trial)

A Protocol Submitted to the Council of the College of Dentistry, University of Baghdad in Partial Fulfillment of Requirements for the Degree of **Master of Science** in Periodontology

By **Sajjad Ahmed Shakir**B.D.S.

Supervised by:
Suzan Ali Salman
MSc

Baghdad-Iraq **2022**, **12**